CLINICAL TRIAL: NCT03486769
Title: Effect of Dual Site-dual Channel Non-invasive Brain Stimulation for Recovery of Motor Function in Stroke Patients
Brief Title: Dual Site-dual Channel Non-invasive Brain Stimulation for Motor Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-08-124-A
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: transcranial direct current stimulation; dual stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dual Stimulation 1 (Experimental): i) anodal stimulation on ipsilesional primary motor cortex and cathodal stimulation on contralesional primary motor cortex, ii) anodal stimulation on ipsilesional premotor cortex and cathodal stimulation on contralesional supraorbital area.
  Interventions: Device: M1 stimulation; Device: PMC stimulation; Behavioral: hand motor task
- Dual Stimulation 2 (Experimental): i) anodal stimulation on ipsilesional primary motor cortex and cathodal stimulation on contralesional primary motor cortex, ii) anodal stimulation on ipsilesional anterior intraparietal sulcus and cathodal stimulation on contralesional supraorbital area.
  Interventions: Device: M1 stimulation; Device: aIPS stimulation; Behavioral: hand motor task
- Single stimulation (Experimental): anodal stimulation on ipsilesional primary motor cortex and cathodal stimulation on contralesional primary motor cortex
  Interventions: Device: M1 stimulation; Behavioral: hand motor task

INTERVENTIONS:
Device: M1 stimulation — stimulating primary motor cortex with anodal transcranial direct current stimulation
  Other Names: primary motor cortex anodal stimulation
Device: PMC stimulation — stimulating premotor cortex with anodal transcranial direct current stimulation
  Other Names: premotor cortex anodal stimulation
  Arms: Dual Stimulation 1
Device: aIPS stimulation — stimulating anterior intraparietal sulcus with anodal transcranial direct current stimulation
  Arms: Dual Stimulation 2
Behavioral: hand motor task — hand motor task for 30 minutes during transcranial direct current stimulation

SUMMARY:
The aim of this study is to investigate the effect of dual site-dual channel non-invasive brain stimulation for recovery of motor function in post stroke patients. Simultaneous dual site-dual channel stimulation was applied by using two sets of transcranial direct current stimulation devices. All subjects will go through three conditions of transcranial direct current stimulation with for 30 minutes. Three conditions are 1) Dual stimulation 1: i) anodal stimulation on ipsilesional primary motor cortex and cathodal stimulation on contralesional primary motor cortex, ii) anodal stimulation on ipsilesional premotor cortex and cathodal stimulation on contralesional supraorbital area. 2) Dual stimulation 2: i) anodal stimulation on ipsilesional primary motor cortex and cathodal stimulation on contralesional primary motor cortex, ii) anodal stimulation on ipsilesional anterior intraparietal sulcus and cathodal stimulation on contralesional supraorbital area. 3) Single stimulation: anodal stimulation on ipsilesional primary motor cortex and cathodal stimulation on contralesional primary motor cortex.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hemiplegic stroke patient
* Fugl Meyer Assessment score between 9 to 84

Exclusion Criteria:

* difficult to understand experimental tasks because of extremely severe cognitive impairment
* history of psychiatric disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Changes in motor evoked potentia | Baseline and after intervention (approximately 2 weeks)
  measure the motor threshold and amplitude of motor evoked potential in first dorsal interosseous muscle.

SECONDARY OUTCOMES:
changes in nine hole peg test | Baseline and after intervention (approximately 2 weeks)
  Nine-Hole Peg Test is used to measure finger dexterity in patients with various neurological diagnoses.
changes in grip and tip pinch strength test | Baseline and after intervention (approximately 2 weeks)
  measure the hand strength (grip and tip pinch)
changes in box and block test | Baseline and after intervention (approximately 2 weeks)
  box and block test measures unilateral gross manual dexterity
Changes in brain activation of resting-state functional MRI | Baseline and after intervention (approximately 2 weeks)
  Neuroplasticity measure
Changes of Cortical activation | Baseline and after intervention (approximately 2 weeks)
  Cortical activation is measured by functional Near-Infrared-Spectroscopy (fNIRS) (NIRScout, NIRx, Germany)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided